CLINICAL TRIAL: NCT04232436
Title: Planned Vaginal Delivery vs Planned Cesarean Delivery in Preterm Twins
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0035
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-01

CONDITIONS: Twin Pregnancy
Keywords: Mode of delivery; Prematurity; Survival at discharge; Survival without severe morbidity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Planned vaginal delivery: Planned vaginal delivery
  Interventions: Other: Survival at discharge; Other: Survival without severe morbidity
- Planned cesarean delivery: Planned cesarean delivery
  Interventions: Other: Survival at discharge; Other: Survival without severe morbidity

INTERVENTIONS:
Other: Survival at discharge — Survival at discharge
Other: Survival without severe morbidity — Survival without severe morbidity (IVH, severe BPD, NEC, ROP)

SUMMARY:
The incidence of twin pregnancies has increased and currently accounts for 1.8% of all deliveries. 47.5% of twins are born prematurely (vs. 6% for singletons) of which 9.9% before 32SA. Caesarean section rates are also higher than for singletons (53.7% vs 19.2%) and 31.8% of caesarean sections are performed before delivery.

The optimal mode of delivery for preterm twins remains controversial. The latest recommendations for clinical practice emphasize that it is not appropriate to recommend one mode of delivery rather than another in the case of twin pregnancies at any term.

In view of all these elements, we wished to carry out a retrospective study at the Montpellier University Hospital in order to compare the neonatal outcome of preterms twins according to their mode of delivery : planned vaginal delivery versus planned cesarean delivery.

ELIGIBILITY:
Inclusion criteria:

* twins born at Montpellier University Hospital
* between 24SA and 32SA+6
* January 2010 to July 2019
* The mothers must have gone into labour spontaneously or after preterm rupture of membranes
* first twin in cephalic presentation

Exclusion criteria:

* twin to twin transfusion syndrome
* monoamniotic pregnancies
* cause of delivery other than preterm labor or preterm rupture of membranes
* lethal malformation
* first twin in breech or transverse presentation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twins born at Montpellier University Hospital between 24SA and 32SA+6
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
survival at discharge and survival | during neonatal hospitalization
  survival at discharge and survival without severe morbidity

SECONDARY OUTCOMES:
survival at 2 years of corrected | during the first two years corrected age
  survival at 2 years of corrected
age without neurosensory impairment | during the first two years corrected age
  age without neurosensory impairment

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC